CLINICAL TRIAL: NCT06286215
Title: Registry of Patients With Plasma Cell Disorders
Acronym: Registry PCD
Status: Not yet recruiting | Type: Observational
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Chutima Kunacheewa, lecturer, Siriraj Hospital
Other Study IDs: 586/2564(IRB2)
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Plasma Cell Disorders
Keywords: registry; plasma cell disorder
MeSH Terms: conditions — Neoplasms, Plasma Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to register patients with plasma cell disorders. The main questions it aims to answer are:

* The incidence of plasma cell disorders both before and after malignancy
* Time to progression of monoclonal gammopathy of undetermined significant (MGUS) or smoldering multiple myeloma (SMM) to light chain amyloidosis or multiple myeloma (MM)
* Progression free survival (PFS)
* overall survival
* factors influencing overall survival, progression-free survival, and time to progression
* Symptoms and signs of the disease during the diagnosis and relapse phases, including the causes of mortality in plasma cell disorder patients.
* genetic characteristics of plasma cell disorder
* cost-effectiveness of treatment in Thailand Participants will be collected the data of baseline diagnosis, treatment, treatment results of all admission and follow-up visits from hospital medical record.

ELIGIBILITY:
Inclusion Criteria:

* Both existing and newly diagnosed patients with plasma cell disorders, including monoclonal gammopathy of undetermined significance, smoldering multiple myeloma, POEMS, light chain amyloidosis, solitary plasmacytoma, and multiple myeloma, according to the diagnostic criteria of the International Myeloma Working Group 2014
* Aged 18 years and above

Exclusion Criteria:

* insufficient data needed for analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: plasma cell disorder patients
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2034-04-01 (Estimated); Study Completion 2035-04-01 (Estimated)

PRIMARY OUTCOMES:
register the plasma cell disorder patients | 10 years
  register the plasma cell disorder patients

SECONDARY OUTCOMES:
incidence of plasma cell disorders | 10 years
  incidence of plasma cell disorders both before and after malignancy
Time to progression | 10 years
  - Time to progression of monoclonal gammopathy of undetermined significant (MGUS) or smoldering multiple myeloma (SMM) to light chain amyloidosis or multiple myeloma (MM)
Progression free survival | 10 years
  Progression free survival
overall survival | 10 years
  overall survival
influencing factors | 10 years
  factors influencing overall survival, progression-free survival, and time to progression
Symptoms and signs | 10 years
  Symptoms and signs of the disease during the diagnosis and relapse phases, including the causes of mortality in plasma cell disorder patients
genetic characteristics | 10 years
  genetic characteristics of plasma cell disorder
cost-effectiveness | 10 years
  cost-effectiveness of treatment in Thailand

IPD SHARING:
Plan to Share IPD: Undecided
Need a consensus from colleagues